CLINICAL TRIAL: NCT02276066
Title: Persistent Inflammation, Immunosuppression and Catabolism Syndrome (PICS): A New Horizon for Surgical Critical Care Subtitle. Kidney Response to Sepsis Affects Angiogenic Balance and Likelihood of CCI and PICS
Brief Title: Kidney Response to Sepsis Affects Angiogenic Balance and Likelihood of CCI and PICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB201400795-N; P50GM111152-01 (NIH)
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Sepsis
Keywords: kidney dysfunction; chronic critical illness; sepsis; Glomerular filtration rate
MeSH Terms: conditions — Sepsis | interventions — Urine Specimen Collection; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhospital group at day 14 (Experimental): This group of sepsis participants remain hospitalized at day 14. GFR assessment is performed at inpatient day 14 and again at 1 year follow up.
  Interventions: Diagnostic Test: GFR by Iohexol; Diagnostic Test: Urine Collection; Diagnostic Test: Blood samples
- Discharged prior to 14 days (Active Comparator): The group of patients were discharged before 14 days. GFR assessment at time of discharge and again at 1 year follow up.
  Interventions: Diagnostic Test: GFR by Iohexol; Diagnostic Test: Urine Collection; Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: GFR by Iohexol — Participants may receive a normal saline dilution of Iohexol 0.5-1 ml given by IV push. Blood or urine will be collected and measured to determine glomerular filtration rate measurements. This test will be repeated in one year.
  Other Names: omnipaque
Diagnostic Test: Urine Collection — Both groups of sepsis participants will have urine collected for at least 4 hours to as long as 24 hours or more. The urine volume determined and a sample sent to the lab for determination of creatinine and urea concentration. This test will be repeated in one year.
Diagnostic Test: Blood samples — Both groups of sepsis participants will provide peripheral blood samples to the research staff. The samples will be sent to the laboratory for serum creatinine results. This test will be repeated in one year.

SUMMARY:
This study investigates the mechanism by which kidney dysfunction perpetuates inflammation, immunosuppression, and catabolism (PICS) in chronic critical illness. The investigators will test the hypothesis that persistent kidney dysfunction in sepsis associated by chronic critical illness contributes to decreased survival through the development of PICS. In chronic critical illness, the persistence of the inflammatory state may lead to capillary rarefication in the kidney causing accelerated chronic kidney disease. Progression of chronic kidney disease during chronic critical illness can drive PICS. Indeed, many of the features of chronic critical illness are consistent with the protein-energy malnutrition and muscle wasting associated with chronic kidney disease. Thus, the kidney can play a contributory role in chronic critical illness and PICS.

DETAILED DESCRIPTION:
The main goal of this project is to measure kidney filtration function at day 14 or the day of discharge from hospital (whichever occurs first), in order to determine the presence and magnitude of persistent kidney dysfunction after sepsis episode and to longitudinally assess further decline of kidney function at one year follow-up. The measure of the glomerular filtration rate (GRF) in patients with chronic critical illness and controls (sepsis patients discharged from ICU before day 14) will be used to determine to what degree of kidney dysfunction contributes to decreased survival and increase in chronic kidney disease at year one after sepsis onset.

GFR assessment will be determined at approximately day 14 or approximately at the day of discharge from the ICU and at the one-year follow-up:

1. Determine GFR by Iohexol clearance and/or
2. Estimated GFR by urea concentration and creatinine clearance
3. Estimated GFR using calculations with serum creatinine

ELIGIBILITY:
Inclusion Criteria:

* Presence in the surgery or trauma ICU
* Age of ≥18 years
* Entrance into our sepsis protocol
* Ability to obtain informed consent.

Exclusion Criteria:

* Expected lifespan of the patient is less than 3 months due to severe pre-existing comorbidities (ex. recurrent, advanced or metastatic cancer)
* Severe traumatic brain injury (evidence of neurologic injury on CT scan and a GCS <8)
* Refractory shock (i.e., patients who die within 12 hours)
* Uncontrollable source of sepsis (e.g., irreversible disease state such as unresectable dead bowel)
* Patient or patient's family are not committed to aggressive management of the patient's condition and/or the patient has a DNR/DNI on file.
* Severe CHF (NY Heart Association Class IV)
* Child-Pugh C liver disease or pre-liver transplant.
* Known HIV infection with CD4 count <200 cells/mm3
* Organ transplant recipient on immunosuppressive agents
* Known pregnancy and mother's that are breastfeeding
* Prisoners
* Institutionalized patients
* Inability to obtain informed consent.
* Chemotherapy or radiotherapy within 30 days prior to sepsis.
* End stage renal disease on admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Segal, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Health at Shands hospital, Gainesville, Florida, United States

REFERENCES:
- [Derived] Loftus TJ, Wu Q, Wang Z, Lysak N, Moore FA, Bihorac A, Efron PA, Mohr AM, Brakenridge SC. Delayed interhospital transfer of critically ill patients with surgical sepsis. J Trauma Acute Care Surg. 2020 Jan;88(1):169-175. doi: 10.1097/TA.0000000000002476. PMID 31856021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 73 subjects enrolled and 41 completed.
Groups:
- Inhospital Group at Day 14: This group of sepsis participants remain hospitalized at day 14.
- Discharged Prior to Hospital Day 14: This group of sepsis participants were discharged prior to day 14.
Period: Overall Study
Arm/Group | Inhospital Group at Day 14 | Discharged Prior to Hospital Day 14
Started | 41 | 32
Completed | 20 | 21
Not Completed | 21 | 11
Not completed — Lost to Follow-up | 21 | 11

BASELINE CHARACTERISTICS:
Groups:
- In Hospital Group at Day 14: This group of sepsis participants remain hospitalized at day 14. A normal saline dilution of Iohexol 0.5-1 ml will be given IV push.
- Discharged From Hospital Prior to Day 14: This group of sepsis participants were discharged prior to day 14 and iohexol determination of GFR was done at time of discharge. A normal saline dilution of Iohexol 0.5-1 ml will be given IV push.
- Total: Total of all reporting groups
Arm/Group | In Hospital Group at Day 14 | Discharged From Hospital Prior to Day 14 | Total
Number analyzed (Participants) | 41 | 32 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 24 | 55
  >=65 years | 10 | 8 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 20 | 13 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 8 | 9
  White | 39 | 24 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 32 | 73
GFR by iohexol [Mean (Standard Deviation); unit: ml/min/1.7m2] — Population: The iohexol could not be performed in many individuals because it was contraindicated or the injection would interfere with patient care.
  ml/min/1.7m2
    number analyzed (Participants) | 20 | 11 | 31
    (all) | 91.5 (46.0) | 88.3 (39.0) | 90.3 (43.0)

OUTCOME MEASURES:

1. Primary Outcome: Delta Curve Between Calculated GFR and GFR Measured by Iohexol at Baseline
Description: The difference between a measured GFR with Iohexol and calculated GFR from creatinine.
Time Frame: For Arm 1 baseline is measured GFR at 14 days inhospital with sepsis or sepsis diagnosis. For Arm 2 baseline is measured GFR at discharge date prior to day 14 of hospitalizaton with sepsis or sepsis diagnosis.
Population: GFR by iohexol and eGFR by CKD epi at baseline. The iohexol could not be performed on many patients because it was contraindicated
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Groups:
- Inhospital Group at Day 14: This group of sepsis participants will remain hospitalized at day 14. A normal saline dilution of Iohexol 0.5-1 ml will be given IV push. Blood or urine will be collected prior to the injection and at approximately 1, 2, 3, and 4 hours after the injection for glomerular filtration rate measurements. This test will be repeated in one year. In addition to or as an option would be to have a timed urine collection to determine clearance of urea and creatinine can be performed instead of the saline dilution of Iohexol 0.5-1 ml and/or an estimated of GFR using serum creatinine and cystatin C measurement using calculations from blood samples.
  Iohexol: Both groups of sepsis participants will receive a normal saline dilution of Iohexol 0.5-1 ml given by IV push. Blood or urine will be collected prior to the injection and at approximately 1, 2, 3, and 4 hours after the injection for glomerular filtration rate measurements. This test will be repeated in one year.
  Urine Collection: Both groups of sepsis participants will have urine collected for at least 4 hours to as long as 24 hours or more. The urine volume determined and a sample sent to the lab for determination of creatinine and urea concentration.
  Blood samples: Both groups of sepsis participants will provide peripheral blood samples to the research staff. The samples will be sent to the laboratory for serum creatinine results.
- Discharged Prior to Day 14 GFR: This group of sepsis participants will remain hospitalized after day 14. A normal saline dilution of Iohexol 0.5-1 ml will be given IV push. The iohexol will be quantified in urine and blood and glomerular filtration rate quantified. This test will be repeated in one year. In addition to or as an option would be to have a timed urine collection to determine clearance of urea and creatinine can be performed instead of the saline dilution of Iohexol 0.5-1 ml and/or an estimated of GFR using serum creatinine and cystatin C measurement using calculations from blood samples.
  Iohexol: Both groups of sepsis participants will receive a normal saline dilution of Iohexol 0.5-1 ml given by IV push. Blood or urine will be collected and measured to determine glomerular filtration rate measurements. This test will be repeated in one year.
  Urine Collection: Both groups of sepsis participants will have urine collected for at least 4 hours to as long as 24 hours or more. The urine volume determined and a sample sent to the lab for determination of creatinine and urea concentration.
  Blood samples: Both groups of sepsis participants will provide peripheral blood samples to the research staff. The samples will be sent to the laboratory for serum creatinine and cystatin C results.
Arm/Group | Inhospital Group at Day 14 | Discharged Prior to Day 14 GFR
Number analyzed (Participants) | 41 | 32
ml/min/1.73m2
  Iohexol GFR: number analyzed (Participants) | 20 | 11
  Iohexol GFR | 91.5 (46.0) | 88.3 (39.0)
  urine collection to determine clearance of urea and creatinine: number analyzed (Participants) | 0 | 0
  eGFR by epi formula | 93.6 (26.6) | 90.0 (28.7)
Statistical Analysis 1: Comparison: Inhospital Group at Day 14 vs Discharged Prior to Day 14 GFR; Test type: Other — We performed a delta analysis, by graphing the difference between the two measurements, we wanted to visually assess the degree of agreement or discrepancy between the two methods. We were looking to evaluate the consistency, accuracy, or bias between different measurement techniques; p < 0.05, Delta analysis

2. Primary Outcome: Delta Curve Between Calculated GFR and GFR Measured by Iohexol at 1 Year Follow-up.
Description: The difference between a measured GFR with Iohexol and calculated GFR from creatinine This was a one-time determination at 1 year follow-up
Time Frame: one year follow up for both arms
Population: The iohexol could not be performed in many individuals because they could not come in to the clinic, would not come into the clinic, or the iohexol injection was contraindicated.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Groups:
- Discharged Prior to 14 Days: These are individuals discharged prior to day 14 inhospital.
Arm/Group | Inhospital Group at Day 14 | Discharged Prior to 14 Days
Number analyzed (Participants) | 3 | 6
mL/min/1.73m2 | 71.4 (38.6) | 58.8 (40.9)

3. Secondary Outcome: Estimated GFR by Serum Creatinine
Description: The correlation between iohexol glomerular filtration rate and estimated glomerular filtration rate using previously validated equation applied to serum creatinine in both groups.
Time Frame: at 14 days inpatient hospitalization or at discharge date prior to day 14 inpatient hospitalization
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Groups:
- Inhospital Group at Day 14: This group of sepsis participants will remain hospitalized after day 14.
- Discharged Prior to Day 14: This group of sepsis participants will be discharged prior day 14.
Arm/Group | Inhospital Group at Day 14 | Discharged Prior to Day 14
Number analyzed (Participants) | 41 | 32
mL/min/1.73m2 | 96.14 (24.77) | 90.0 (28.7)

4. Secondary Outcome: Estimated GFR by Serum Creatinine
Description: as for outcome 3
Time Frame: at 1 year follow-up
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Groups:
- Inhospital Group at Day 14: This group of sepsis participants will remain hospitalized at day 14.
- Discharged Prior to Day 14: Subjects discharged prior to hospital day 14
Arm/Group | Inhospital Group at Day 14 | Discharged Prior to Day 14
Number analyzed (Participants) | 20 | 21
ml/min/1.73m2 | 83.0 (25.3) | 83.2 (29.2)

5. Secondary Outcome: Calculated GFR by Urea Concentration and Creatinine Clearance
Description: The urine will be collected for at least 4 hours to as long as 24 hours or more. The urine volume determined and a sample sent to the lab for determination of creatinine and urea concentration
Time Frame: at 14 days inpatient hospitalization or at discharge date prior to day 14 inpatient hospitalization
Population: this outcome measure was not performed due to lack of funding prior to initiation of study
Groups:
- Discharged Prior to Day 14: This group of sepsis participants will be discharged prior to hospitalization day 14.
Arm/Group | Inhospital Group at Day 14 | Discharged Prior to Day 14
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Calculated GFR by Urea Concentration and Creatinine Clearance
Description: as for outcome 5
Time Frame: at one year follow-up
Population: this outcome measure not performed due to funding cuts prior to initiation of study
Groups:
- Discharged Prior to Hospital Day 14: This group of sepsis participants were discharged prior to hospitalization day 14.
Arm/Group | Inhospital Group at Day 14 | Discharged Prior to Hospital Day 14
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for an entire year after consent was signed. We report all adverse events for all individuals enrolled in this trial. No adverse events were related to this trial or the larger trial, but the study involved critically ill subjects, so there were a lot of serious adverse events. Thus all adverse events that occurred after the subject signed consent and for the next 365 days are reported.
Description: We report all adverse events for all individuals enrolled in this trial.
Groups:
- Inhospital Group at Day 14: This group of sepsis participants will remain hospitalized at day 14. GFR assessment at inpatient day 14 and again at 1 year follow up
- Discharged From Hospital Prior to Day 14: The group discharged before 14 days hospitalizaton. GFR assessment at discharge and again at 1 year follow-up
Arm/Group | Inhospital Group at Day 14 | Discharged From Hospital Prior to Day 14
All-Cause Mortality (participants affected / at risk) | 6/41 | 1/32
Serious Adverse Events (participants affected / at risk) | 24/41 | 15/32
Other Adverse Events (participants affected / at risk) | 0/41 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhospital Group at Day 14 (N=41) | Discharged From Hospital Prior to Day 14 (N=32)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3) — readmitted with a chief complaint of abdominal pain
colostomy reversal (Gastrointestinal disorders) | 1 (1) | 0 (0) — Readmission for colostomy reversal
Blood Transfusion (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Readmission for wound care (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Readmission for pacemaker implant (Cardiac disorders) | 0 (0) | 1 (1)
Readmission for planned angiogram (Vascular disorders) | 0 (0) | 1 (1)
Esophagael surgery (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Sepsis (General disorders) | 1 (1) | 0 (0)
Altered Mental Status (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 6 (6) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 0 (0) | 2 (2)
cholecystectomy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pancreatic Surgery (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
C. Diff infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT02276066/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT02276066/ICF_001.pdf